CLINICAL TRIAL: NCT04413617
Title: A 24-WEEK RANDOMIZED, DOUBLE-BLIND, PARALLEL GROUP, ACTIVE COMPARATOR, MULTICENTER STUDY TO ASSESS THE EFFICACY AND SAFETY OF PF-06650833, PF-06651600 (RITLECITINIB) AND TOFACITINIB ALONE AND IN COMBINATION IN PARTICIPANTS WITH MODERATELY-SEVERELY ACTIVE RHEUMATOID ARTHRITIS WITH AN INADEQUATE RESPONSE TO METHOTREXATE
Brief Title: TO ASSESS THE EFFICACY AND SAFETY OF PF-06650833, PF-06651600, AND TOFACITINIB ALONE AND IN COMBINATION IN PARTICIPANTS WITH ACTIVE RHEUMATOID ARTHRITIS WITH AN INADEQUATE RESPONSE TO METHOTREXATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7921023; 2019-002676-14 (EudraCT Number)
Record Dates: First submitted 2020-05-19; First posted 2020-06-04 (Actual); Results first posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — 1-(((2S,3S,4S)-3-ethyl-4-fluoro-5-oxopyrrolidin-2-yl)methoxy)-7-methoxyisoquinoline-6-carboxamide; PF-06651600; tofacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- PF-06650833 + tofacitinib (Experimental)
  Interventions: Drug: PF-06650833; Drug: Tofacitinib
- PF-06650833 + PF-06651600 (Experimental)
  Interventions: Drug: PF-06650833; Drug: PF-06651600
- PF-06650833 (Experimental)
  Interventions: Drug: PF-06650833
- PF-06651600 (Experimental)
  Interventions: Drug: PF-06651600
- Tofacitinib (Experimental)
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: PF-06650833 — 400 mg
  Arms: PF-06650833; PF-06650833 + PF-06651600; PF-06650833 + tofacitinib
Drug: PF-06651600 — 100 mg
  Arms: PF-06650833 + PF-06651600; PF-06651600
Drug: Tofacitinib — 11 mg
  Arms: PF-06650833 + tofacitinib; Tofacitinib

SUMMARY:
Dual objectives of increased efficacy compared to currently available SoC RA drugs and maintaining a favourable benefit - risk relationship.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants between the ages of 18 and 70 years.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Diagnosis of RA and meeting the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria for RA with a Total Score ≥6/10.
* The participant has active disease at both Screening and Randomization, as defined by both: ≥6 joints tender or painful on motion, AND ≥6 joints swollen; and fulfills 1 of the following 2 criteria: High sensitivity C reactive protein (hsCRP) >7 mg/L at Screening (Visit 1) as performed by the central laboratory OR Erythrocyte sedimentation rate (ESR) (Westergren method) >28 mm h.

Exclusion Criteria:

* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or IP administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Participants with a known immunodeficiency disorder or a first degree relative with a hereditary immunodeficiency.
* Participants with any active or latent infections.
* Participants with positive hepatitis B surface antigen (HBsAg).
* Participants with positive HCV Ab tests will be reflex tested for HCV ribonucleic acid (HCV RNA).
* Any history of either untreated or inadequately treated latent or active tuberculosis (TB) infection, current treatment for active or latent TB infection or evidence of currently active TB,
* History of a major organ transplant (eg, heart, lung, kidney and liver) or hematopoietic stem cell/marrow transplant.
* History of severe allergic or anaphylactoid reaction to kinase inhibitors, or corticosteroid preparations.
* Known history of diverticulitis or symptomatic diverticulosis, perineal abscess or fistulae.
* Participants with malignancy or history of malignancy (including lymphoma, leukemia, or lymphoproliferative disease).
* Pre-existing chronic autoimmune disease (eg, inflammatory bowel disease, systemic lupus erythematosus, moderate-severe atopic dermatitis, dermatomyositis) other than RA. Secondary Sjogren's Syndrome (due to RA) may be included.
* Participants with fibromyalgia will be excluded.
* Previous treatment with total lymphoid irradiation.
* Participants with an oral, tympanic, or temporal temperature of 38°C (100.4°F) or higher at baseline.
* Participants may not receive any live/attenuated vaccine from 30 days prior to randomization during the course of the study, or for 30 days after the last dose of study medication. Participants who have current routine household contact with children who have received varicella or oral polio vaccine within 2 months of first study dose are also excluded.
* History of any lymphoproliferative disorder.
* Have hearing loss with progression over the previous 5 years, sudden hearing loss, or middle or inner ear disease.
* History of any prior deep vein thrombosis (DVT) or pulmonary embolism [PE].
* Recent (within 6 months of screening) myocardial infarction, coronary revascularization, or percutaneous angioplasty with or without placement of a coronary artery stent; acute coronary syndrome; chronic uncompensated heart failure or New York Heart Association Functional Class III or IV; left ventricular assist devices; implanted defibrillators.
* Current severe chronic renal insufficiency or renal failure as defined by persistent (on repeated measurements) eGFR <60 mL/min per 1.73 m2 based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) calculation.
* Any known coagulopathy or hypercoagulant syndrome.
* Presence of any of the following laboratory abnormalities at screening or within the 3 months prior to first study dose:

Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels ≥1.5 x the upper limit of normal (ULN); Participants with a history of Gilbert's syndrome may have a direct bilirubin measured and would be eligible for this study provided the direct bilirubin is ≤ ULN and other liver function assessments are normal; Absolute neutrophil count of <1.5 x 109/L (<1500/mm3). Participants with cyclic (benign ethnic) neutropenia will be excluded; Absolute lymphocyte count of <0.5 x 109/L (<500/mm3); Absolute white blood cell (WBC) count of <3.0 x 109/L (<3000/mm3); Hemoglobin <9.0 g/dL (90 g/L); Platelet count ≤100 x 109/L (100,000 cells/mm3) or ≥1000 x 109/L (1,000,000 cells/mm3); Thrombocytopenia, as defined by a platelet count <100 x 109/L (<100,000/mm3) at screening visit or within the 3 months prior to first study dose. [Screening laboratory tests with abnormal results may be repeated once to confirm abnormal results. If results return to normal protocol acceptable limits within the 4-week screening period, the participant may enter the study].

- Grade 3 or greater laboratory abnormality based on the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 toxicity scale, except for the following that are allowed: Grade 3 prothrombin time (PT) secondary to warfarin treatment; Grade 3 partial thromboplastin time (PTT) due to lupus anticoagulant and not related to liver disease or anti-coagulant therapy.

* Participants previously treated with a biologic DMARD (except for up to 25% of participants who may have been treated with 1, and only 1 prior TNF inhibitor) or any other recent DMARD treatment (eg, a JAK inhibitor), or participants currently treated with any other prohibited medications will be excluded.
* Prior use of tofacitinib or other JAK inhibitor in the context of a clinical trial is excluded. Concomitant use of tofacitinib (other than as prescribed by the randomization scheme) or other JAK inhibitor is prohibited.
* Participants who have previously been treated with other, non-TNFa inhibiting biologic DMARDs [including, abatacept (Orencia®), tocilizumab (Actemra®), Sarilumab (Kevzara®), anakinra (Kineret®), rituximab (Rituxan®) or other selective B lymphocyte depleting agents, or other lymphocyte depleting agents/therapies (such as alemtuzab [CamPath®], natalizumab (Tysabri®), alkylating agents [eg, cyclophosphamide or chlorambucil], total lymphoid irradiation) are excluded from participation in the study.
* Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of IP used in this study (whichever is longer).
* Any 12-lead electrocardiogram (ECG) performed prior to randomization that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (143):
- Bulgaria (12):
  - ,,UMHAT - Georgi Stranski" EAD, Pleven
  - Medical Diagnostic Laboratory Rusev EOOD, Plovdiv
  - MHAT Plovdiv AD, Plovdiv
  - DCC Sveti Georgi EOOD, Plovdiv
  - Independent Medical Diagnostic Laboratory Mediscan EOOD, Plovdiv
  - "Medical Center-Teodora" EOOD, Rousse
  - UMHAT "Kanev" AD, Rousse
  - Medical Center "Spectar" OOD, Sofia
  - MHAT "Lyulin" EAD, Sofia
  - "DCC 17 - Sofia" EOOD, Sofia
  - Medical Center "N.I. Pirogov" EOOD, Sofia
  - UMHAT "Sveti Ivan Rilski" EAD, Sofia
- Canada (2):
  - Manitoba Clinic, Winnipeg, Manitoba
  - Centre de Rhumatologie de l'Est du Quebec (CREQ), Rimouski, Quebec
- Chile (6):
  - Centro Radiologico San Vicente de Paul, Santiago, Santiago Metropolitan
  - CTR Estudios, Santiago, Santiago Metropolitan
  - Enroll SpA, Santiago, Santiago Metropolitan
  - Centro Radiologico Plaza Baquedano, Santiago, Santiago Metropolitan
  - IMARED, Santiago, Santiago Metropolitan
  - Centro de Estudios Reumatologicos (CER), Santiago, Santiago Metropolitan
- Czechia (16):
  - CCR Czech a.s., Pardubice, Vychodocesky KRAJ
  - REVMACLINIC s.r.o., Brno
  - Revmacentrum MUDr. Mostera, s.r.o., Brno
  - HV Medical s.r.o., ORL ambulance pro deti a dospele, Brno
  - MRI Lekarsky servis s.r.o., Havířov
  - CCR Ostrava, s.r.o., Ostrava
  - Vesalion s.r.o., Ostrava
  - Mestka nemocnice Ostrava, Ostrava
  - Poliklinika AMO - Audiologie, Ostrava-Kunčice
  - ORL - sluchadla s.r.o., Pardubice
  - Poliklinika Vektor, Pardubice
  - Revmatologicky ustav, Prague
  - Thomayerova nemocnice, Prague
  - ORL ambulance, Uherské Hradiště
  - Uherskohradistska nemocnice, a.s., Uherské Hradiště
  - Medical Plus s.r.o., Uherské Hradiště
- Georgia (5):
  - JSC "Evex Hospitals", Tbilisi
  - LTD "Cardioclinic - Digomi Medical Center", Tbilisi
  - LTD "Institute of Clinical Cardiology", Tbilisi
  - LTD "MediClub Georgia", Tbilisi
  - LTD "Multi-Profile Clinic Consilium Medulla", Tbilisi
- Hungary (23):
  - Trial Pharma Kft., Békéscsaba
  - Vasutegeszsegugyi Nonprofit Kozhasznu Tarsasag, Békéscsaba
  - Betegapolo Irgalmasrend Budai Irgalmasrendi Korhaz, Budapest
  - Mammut Egeszsegkozpont, Ful-orr- gegeszet, Budapest
  - Budai Irgalmasrendi Korhaz, Budapest
  - Revita Reumatologiai Rendelo, Budapest
  - Qualiclinic Kft., Budapest
  - Affidea Magyarorszag Kft., Budapest
  - Affidea Magyarország Kft. Bank Center Központ, Budapest
  - Magyar Honvédség Egészségügyi Központ, Budapest
  - Affidea Magyarorszag Kft. Vaci Greens Egeszsegkozpont, Budapest
  - Mediszintech Audiologia Kft., Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - Sanitas Diagnosztikai es Rehabilitacios Kozpont, Gyula
  - Pest Megyei Flór Ferenc Kórház Fül- Orr- Gégészet és Gyermek Fül-Orr-Gégészet, Kistarcsa
  - Pest Megyei Flór Ferenc Kórház Reumatológiai es Fizioterápiás Osztály, Kistarcsa
  - Huniko Kereskedelmi és Egészségügyi Szolgáltató Kft., Miskolc
  - Szegedi Tudomanyegyetem Reumatologiai Klinika, Szeged
  - Szegedi Tudomanyegyetem, Szeged
  - Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
  - Csolnoky Ferenc Korhaz, Ful- Orr- Gegeszeti Osztaly, Veszprém
  - VITAL MEDICAL CENTER (VITÁL-MEDICINA Kft.), Veszprém
- Poland (39):
  - Podlaskie Centrum Sluchu i Mowy Sluchmed, Bialystok
  - Nzoz Zdrowie Osteo-Medic, Bialystok
  - Lar-Med, Bialystok
  - NZOZ Kendron, Bialystok
  - Tomma Diagnostyka obrazowa, Bialystok
  - ClinicMed Daniluk, Nowak Sp. J., Bialystok
  - Nzoz McD Voxel, Bydgoszcz
  - Klinika Foniatrii i Audiologii, Szpital Uniwersytecki Nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Klinika Reumatologii i Ukladowych Chorob Tkanki Lacznej, Bydgoszcz
  - Centrum Medyczne Pratia Gdynia, Gdynia
  - Portowy Zaklad Opieki Zdrowotnej Sp. z o.o., Gdynia
  - Centrum Medyczne Enel-Med., Oddzial Alfa Plaza - Gdynia, Gdynia
  - MCBK, Grodzisk Mazowiecki
  - Samodzielny Publiczny Specjalistyczny Szpital Zachodni im. sw. Jana Pawla II, Grodzisk Mazowiecki
  - Malopolskie Badania Kliniczne, Krakow
  - LUX MED., Krakow
  - Centrum Badan Klinicznych JCI, Krakow
  - Centrum medyczne PLEJADY, Krakow
  - LUXMED, Krakow
  - Pratia MCM Krakow, Krakow
  - Centrum Medycyny Profilaktycznej Sp. z o. o., Krakow
  - Centrum Medyczne iMed24, Krakow
  - FONMED, Nowa Sól
  - Twoja Przychodnia - Centrum Medyczne Nowa Sol, Nowa Sól
  - LIVMED Sp. z.o.o., Nowy Tomyśl
  - Ai Centrum Medyczne, Poznan
  - Tomma Diagnostyka Obrazowa S.A., Poznan
  - GEERS Dobry Sluch, Poznan
  - Prywatna Praktyka Lekarska Prof. dr hab. med. Pawel Hrycaj, Poznan
  - Pracownia Rezonansu Magnetycznego i RTG, Poznan
  - Centrum Mowy i Sluchu Medincus, Warsaw
  - Rex Medica Sport, Warsaw
  - Medycyna Kliniczna, Warsaw
  - Tomma Diagnostyka Obrazowa, Warsaw
  - "MTZ CLINICAL RESEARCH" Spolka z ograniczona odpowiedzialnoscia, Warsaw
  - "Reumatika - Centrum Reumatologii" NZOZ, Warsaw
  - ArtAna Anna Piotrowska, Warsaw
  - Spoldzielnia Pracy Specjalistow Rentgenologow im. prof. W. Zawadowskiego, Warsaw
  - Szpital LUX MED, Warsaw
- Slovakia (23):
  - Dermatovenerologicka ambulancia, Bratislava
  - ROMJAN, s.r.o., Bratislava
  - ORL ambulancia RHINO s.r.o., Bratislava
  - Klinika dermatovenerologie UNLP, Košice
  - ARTROMAC n. o., Košice
  - Oddelenie radiodiagnostiky a zobrazovacich metod, UNLP, Košice
  - Poliklinika Terasa s.r.o., Košice
  - Dermabene, s.r.o, Martin
  - MEDMAN, s. r. o.,, Martin
  - ORL ML, s.r.o, Martin
  - Jessenius - Diagnosticke centrum, Nitra
  - Otorinolaryngologicka ambulancia MUDr. Olga Salgova, Partizánske
  - PARDERM, s. r. o., Dermatovenerologicka ambulancia, Partizánske
  - REUMACENTRUM s.r.o., Partizánske
  - MEDICENTRUM Piestany, s.r.o., Piešťany
  - Narodny ustav reumatickych chorob, Piešťany
  - Nemocnica Alexandra Wintera n.o., Piešťany
  - Vseobecna nemocnica Rimavska Sobota, Rimavská Sobota
  - AZIMED-ORL s.r.o., Rimavská Sobota
  - Dg.s.r.o. - Diagnosticke- centrum, Rimavská Sobota
  - REUMEX s.r.o., Rimavská Sobota
  - Spinn, s.r.o., Ružomberok
  - Zdravomak s.r.o. Topoľčany, Topoľčany
- Spain (6):
  - Clinica Gaias - Santiago, Santiago de Compostela, A Coruna
  - Grupo Hospitalario La Rosaleda - Hospital Nuestra Senora de la Esperanza, Santiago de Compostela, A Coruna
  - Hospital General Universitario de Elche, Elche, Alicante
  - Clinica Sagrada Familia, Barcelona
  - Hospital Clinico Universitario Santiago de Compostela, Santiago de Compostela
  - Hospital Quironsalud Infanta Luisa, Seville
- Ukraine (11):
  - Communal non-profit enterprise "Chernihiv Regional Hospital" of Chernihiv Regional Council, Chernihiv
  - Communal Non-commercial Enterprise of Kharkiv Regional Council, Kharkiv
  - Medical сепtег of "Medical Clinic "Blagomed" LLC, Kyiv
  - Medical Center 'Ok!Clinic+' of International Institute of Clinical Research LLC, Kyiv
  - Communal non-profit enterprise "Kyiv City Clinical Hospital #3" of executive body of Kyiv, Kyiv
  - Limited Liability Company "Medical Centre "Consilium Medical", Kyiv
  - "Revmocenter" LLC, Kyiv
  - Clinic of the State Institution "DF Chebotaryov Institute of Gerontology of the NAMS of Ukraine", Kyiv
  - Communal Non-Commercial Enterprise "Odesa Regional Clinical Hospital" of Odesa Regional Council, Odesa
  - Comunal Enterprise "Poltava Regional Clinical Hospital n. a. M.S. Sklifosovskogo of Poltava, Poltava
  - LLC "Modern Clinic", Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7921023

RESULTS

PARTICIPANT FLOW:
Groups:
- Tofacitinib 11mg MR: Participants received tofacitinib 11mg as modified release (MR) tablets once daily (QD).
- PF-06651600 100mg: Participants received PF-06651600 100mg tablets QD.
- PF-06650833 400mg MR: Participants received PF-06650833 400mg as MR tablets QD.
- PF-06650833 400mg MR + Tofacitinib 11mg MR: Participants received PF-06650833 400mg MR tablets coadministered with tofacitinib 11mg MR tablets QD.
- PF-06650833 400mg MR + PF-06651600 100mg: Participants received PF-06650833 400mg MR tablets coadministered with PF-06651600 100mg tablets QD.
Period: Overall Study
Arm/Group | Tofacitinib 11mg MR | PF-06651600 100mg | PF-06650833 400mg MR | PF-06650833 400mg MR + Tofacitinib 11mg MR | PF-06650833 400mg MR + PF-06651600 100mg
Started | 102 | 77 | 77 | 103 | 101
Completed | 95 | 71 | 73 | 95 | 96
Not Completed | 7 | 6 | 4 | 8 | 5
Not completed — Refused to come for FU visit and was contacted by phone | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 1
Not completed — Lack of Efficacy | 2 | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 4 | 2 | 5 | 3
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 1
Not completed — COVID-19 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the intervention they actually received.
Groups:
- Tofacitinib 11mg MR: Participants received tofacitinib 11mg MR tablets QD.
- Total: Total of all reporting groups
Arm/Group | Tofacitinib 11mg MR | PF-06651600 100mg | PF-06650833 400mg MR | PF-06650833 400mg MR + Tofacitinib 11mg MR | PF-06650833 400mg MR + PF-06651600 100mg | Total
Number analyzed (Participants) | 102 | 77 | 77 | 103 | 101 | 460
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.2 (10.63) | 52.8 (10.90) | 53.6 (9.87) | 54.0 (10.41) | 53.0 (10.40) | 52.9 (10.46)
Age, Customized [Count of Participants; unit: Participants]
  18-44 | 25 | 17 | 11 | 19 | 21 | 93
  45-64 | 68 | 49 | 56 | 71 | 66 | 310
  >=65 | 9 | 11 | 10 | 13 | 14 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 62 | 61 | 78 | 73 | 356
  Male | 20 | 15 | 16 | 25 | 28 | 104
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 101 | 76 | 77 | 102 | 101 | 457
  Asian | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1
  Multiracial | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) in Disease Activity Score (DAS)28-C Reactive Protein (CRP) at Week 12
Description: DAS28 is a measure based on assessment of 28 joints for tenderness and swelling (tender and swollen joint counts). Disease Activity Score 28-C reactive protein (DAS28-CRP) is derived using differential weighting given to 4 components: tender joint count (range: 0-28), swollen joint count (range: 0-28), patient global assessment (recorded on a visual analog scale [VAS] scale of 0-100 mm), and CRP (milligram per liter). DAS28-CRP score ranges from 0 to 9.4. The lower the DAS28-CRP score is, the better the participant has response (remission = score<2.6, low disease activity = score≤3.2). A negative value in change from BL indicates an improvement. Mixed Model Repeated Measures was used for statistical analysis, which used the change from BL of DAS28-CRP as an outcome and treatment, scheduled study visit, BL value of DAS28-CRP, treatment by visit interaction and BL by visit interaction as fixed effects. The model used the unstructured covariance matrix.
Time Frame: BL (defined as the last non-missing measurement collected prior to the first administration of study drug on Day 1), Week 12
Population: The primary efficacy endpoint used Modified Intent to Treat (mITT) data set, which included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the randomized intervention. Participants with non-missing data at a given visit were included.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Groups:
- PF-06650833 400mg MR + Tofacitinib 11mg MR: Participants who received PF-06650833 400mg MR coadministered with tofacitinib 11mg MR
- PF-06650833 400mg MR + PF-06651600 100mg: Participants who received PF-06650833 400mg MR coadministered with PF-06651600 100mg
- Tofacitinib 11mg MR: Participants who received tofacitinib 11mg MR
- PF-06651600 100mg: Participants who received PF-06651600 100mg
- PF-06650833 400mg MR: Participants who received PF-06650833 400mg MR
Arm/Group | PF-06650833 400mg MR + Tofacitinib 11mg MR | PF-06650833 400mg MR + PF-06651600 100mg | Tofacitinib 11mg MR | PF-06651600 100mg | PF-06650833 400mg MR
Number analyzed (Participants) | 96 | 93 | 96 | 69 | 71
Units on a scale | -2.65 [-2.84 to -2.46] | -2.35 [-2.54 to -2.15] | -2.30 [-2.49 to -2.11] | -2.20 [-2.43 to -1.98] | -1.82 [-2.04 to -1.60]
Statistical Analysis 1: Comparison: PF-06650833 400mg MR + Tofacitinib 11mg MR vs Tofacitinib 11mg MR; The primary clinical hypothesis is that mean decrease at Week 12 in DAS28-CRP score in one or both combo arms exceeds the mean decrease in the reference (tofacitinib) treatment arm, regardless of occurrence of intercurrent events. The null hypothesis is that the mean decrease in DAS28-CRP score at Week 12 is identical in the control (tofacitinib arm) and combination arms; Test type: Superiority; p = 0.0158, Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.35, 90% CI 2-sided [-0.62 to -0.08], Standard Error of Mean 0.163
Statistical Analysis 2: Comparison: PF-06650833 400mg MR + PF-06651600 100mg vs Tofacitinib 11mg MR; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3933, Mixed Model Repeated Measures; Mean Difference (Final Values) = -0.04, 90% CI 2-sided [-0.32 to 0.23], Standard Error of Mean 0.164

2. Secondary Outcome: DAS28-CRP Remission (<2.6) Rates at Week 24
Description: DAS28-CRP is derived using differential weighting given to 4 components: tender joint count, swollen joint count, patient global assessment, and CRP. Remission is defined as DAS28-CRP score <2.6. Remission rate = the number of responders (who had remission) / (number of responders + non-responders + non-responder assigned by non-responder imputation [NRI] after removal of missingness due to COVID-19 and missing components at a given visit)
Time Frame: Week 24
Population: The NRI data set included responders, non-responders, and non-responder assigned by NRI after removal of missingness due to COVID-19 and missing components at a given visit.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-06650833 400mg MR + Tofacitinib 11mg MR | PF-06650833 400mg MR + PF-06651600 100mg | Tofacitinib 11mg MR | PF-06651600 100mg | PF-06650833 400mg MR
Number analyzed (Participants) | 103 | 99 | 100 | 76 | 76
Percentage of participants | 40.8 [32.6 to 48.7] | 31.3 [24.1 to 39.8] | 24.0 [17.1 to 31.8] | 22.4 [14.8 to 31.3] | 11.8 [6.7 to 19.3]

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs), and Withdrawals Due to TEAEs
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical study subject, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious AE (SAE) was defined as any untoward medical occurrence that, at any dose: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent disability/incapacity; was a congenital anomaly/birth defect; or other serious situations such as important medical events. TEAEs were events between first dose of study drug and up to follow-up visit that were absent before treatment or that worsened after treatment. AEs presented below were TEAEs. The investigator was required to use clinical judgment to assess the potential relationship between investigational product and each AE, to define an treatment-related AE.
Time Frame: From first dose of study intervention (Day 1) to Week 28
Population: The safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 11mg MR | PF-06651600 100mg | PF-06650833 400mg MR | PF-06650833 400mg MR + Tofacitinib 11mg MR | PF-06650833 400mg MR + PF-06651600 100mg
Number analyzed (Participants) | 102 | 77 | 77 | 103 | 101
Participants
  All-causality TEAEs | 60 | 42 | 38 | 51 | 55
  Treatment-related TEAEs | 15 | 17 | 13 | 20 | 25
  All-causality TESAEs | 3 | 3 | 3 | 0 | 1
  Treatment-related TESAEs | 0 | 0 | 0 | 0 | 0
  Discontinuation from study due to all-causality TEAEs | 2 | 0 | 0 | 1 | 1
  Discontinuation from study due to treatment-related TEAEs | 1 | 0 | 0 | 1 | 0
  Study drug withdrawal due to all-causality TEAEs but continued study | 0 | 6 | 6 | 4 | 6
  Study drug withdrawal due to treatment-related TEAEs but continued study | 0 | 4 | 4 | 3 | 4

4. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities (Hematology and Chemistry, Without Regard to Baseline Abnormality)
Description: Clinical laboratory abnormality was determined at the investigator's discretion.
Time Frame: From BL to Week 28
Population: The analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants with evaluable laboratory values were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 11mg MR | PF-06651600 100mg | PF-06650833 400mg MR | PF-06650833 400mg MR + Tofacitinib 11mg MR | PF-06650833 400mg MR + PF-06651600 100mg
Number analyzed (Participants) | 101 | 77 | 77 | 102 | 101
Participants
  Hematology: Hemoglobin (gram per deciliter [g/dL]) <0.8x lower limit of normal (LLN): number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Hematology: Hemoglobin (gram per deciliter [g/dL]) <0.8x lower limit of normal (LLN) | 2 | 2 | 0 | 2 | 2
  Erythrocytes (10^6/millimeter^3 [10^6/mm^3]) <0.8x LLN: number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Erythrocytes (10^6/millimeter^3 [10^6/mm^3]) <0.8x LLN | 0 | 2 | 0 | 0 | 0
  Erythrocyte (Ery.) Mean Corpuscular Volume (micrometer^3 [um^3]) <0.9x LLN: number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Erythrocyte (Ery.) Mean Corpuscular Volume (micrometer^3 [um^3]) <0.9x LLN | 3 | 2 | 0 | 2 | 0
  Ery. Mean Corpuscular Volume (um^3) >1.1x upper limit of normal (ULN): number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Ery. Mean Corpuscular Volume (um^3) >1.1x upper limit of normal (ULN) | 4 | 3 | 4 | 3 | 4
  Ery. Mean Corpuscular Hemoglobin (picogram/cell [pg/cell]) <0.9x LLN: number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Ery. Mean Corpuscular Hemoglobin (picogram/cell [pg/cell]) <0.9x LLN | 8 | 5 | 3 | 7 | 4
  Ery. Mean Corpuscular Hemoglobin (HGB) Concentration (g/dL) <0.9x LLN: number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Ery. Mean Corpuscular Hemoglobin (HGB) Concentration (g/dL) <0.9x LLN | 8 | 6 | 12 | 10 | 4
  Platelets (10^3/mm^3) >1.75xULN: number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Platelets (10^3/mm^3) >1.75xULN | 0 | 0 | 0 | 1 | 0
  Reticulocytes/Erythrocytes (%) >1.5x ULN: number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Reticulocytes/Erythrocytes (%) >1.5x ULN | 2 | 1 | 2 | 1 | 1
  Leukocytes (10^3/mm^3) <0.6x LLN: number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Leukocytes (10^3/mm^3) <0.6x LLN | 0 | 1 | 0 | 0 | 1
  Leukocytes (10^3/mm^3) >1.5x ULN: number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Leukocytes (10^3/mm^3) >1.5x ULN | 2 | 2 | 1 | 1 | 3
  Lymphocytes (10^3/mm^3) <0.8x LLN: number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Lymphocytes (10^3/mm^3) <0.8x LLN | 7 | 16 | 3 | 6 | 13
  Lymphocytes (10^3/mm^3) >1.2x ULN: number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Lymphocytes (10^3/mm^3) >1.2x ULN | 3 | 2 | 1 | 1 | 2
  Lymphocytes/Leukocytes (%) <0.8x LLN: number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Lymphocytes/Leukocytes (%) <0.8x LLN | 6 | 11 | 9 | 6 | 10
  Lymphocytes/Leukocytes (%) >1.2x ULN: number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Lymphocytes/Leukocytes (%) >1.2x ULN | 1 | 1 | 1 | 5 | 3
  Neutrophils (10^3/mm^3) <0.8x LLN: number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Neutrophils (10^3/mm^3) <0.8x LLN | 2 | 2 | 3 | 5 | 4
  Neutrophils (10^3/mm^3) >1.2x ULN: number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Neutrophils (10^3/mm^3) >1.2x ULN | 11 | 16 | 8 | 5 | 14
  Neutrophils/Leukocytes (%) <0.8x LLN: number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Neutrophils/Leukocytes (%) <0.8x LLN | 1 | 0 | 0 | 2 | 1
  Neutrophils/Leukocytes (%) >1.2x ULN: number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Neutrophils/Leukocytes (%) >1.2x ULN | 5 | 9 | 6 | 3 | 7
  Basophils (10^3/mm^3) >1.2x ULN: number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Basophils (10^3/mm^3) >1.2x ULN | 0 | 0 | 1 | 1 | 0
  Eosinophils (10^3/mm^3) >1.2x ULN: number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Eosinophils (10^3/mm^3) >1.2x ULN | 0 | 0 | 3 | 1 | 0
  Eosinophils/Leukocytes (%) >1.2x ULN: number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Eosinophils/Leukocytes (%) >1.2x ULN | 1 | 0 | 5 | 4 | 1
  Monocytes (10^3/mm^3) >1.2x ULN: number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Monocytes (10^3/mm^3) >1.2x ULN | 2 | 1 | 1 | 0 | 2
  Monocytes/Leukocytes (%) >1.2x ULN: number analyzed (Participants) | 101 | 77 | 77 | 101 | 101
  Monocytes/Leukocytes (%) >1.2x ULN | 8 | 12 | 6 | 11 | 17
  Activated Partial Thromboplastin Time (second [sec]) >1.1x ULN | 9 | 9 | 9 | 10 | 10
  Prothrombin Time (sec) >1.1x ULN | 7 | 6 | 6 | 2 | 9
  Erythrocyte Sedimentation Rate (millimeter per hour [mm/hr]) >1.5x ULN | 72 | 59 | 58 | 71 | 63
  Clinical Chemistry: Bilirubin (milligram per deciliter [mg/dL]) >1.5x ULN | 2 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase (AST) (unit per liter [U/L]) >3.0x ULN | 0 | 0 | 2 | 1 | 0
  Alanine Aminotransferase (ALT) (U/L) >3.0x ULN | 0 | 1 | 7 | 2 | 0
  Urea Nitrogen (mg/dL) >1.3x ULN | 4 | 1 | 5 | 4 | 2
  Creatinine (mg/dL) >1.3x ULN | 0 | 0 | 0 | 1 | 0
  Urate (mg/dL) >1.2x ULN | 3 | 2 | 2 | 4 | 1
  Cholesterol (mg/dL) >1.3x ULN: number analyzed (Participants) | 94 | 71 | 73 | 100 | 91
  Cholesterol (mg/dL) >1.3x ULN | 22 | 13 | 10 | 24 | 20
  High-Density Lipoprotein (HDL) Cholesterol (mg/dL) <0.8x LLN: number analyzed (Participants) | 94 | 70 | 69 | 98 | 90
  High-Density Lipoprotein (HDL) Cholesterol (mg/dL) <0.8x LLN | 1 | 3 | 1 | 0 | 1
  Low-Density Lipoprotein (LDL) Cholesterol (mg/dL) >1.2x ULN: number analyzed (Participants) | 92 | 70 | 68 | 98 | 88
  Low-Density Lipoprotein (LDL) Cholesterol (mg/dL) >1.2x ULN | 9 | 5 | 1 | 5 | 8
  Sodium (milliequivalent per liter [mEq/L]) <0.95x LLN | 0 | 1 | 0 | 0 | 0
  Potassium (mEq/L) <0.9x LLN | 0 | 1 | 2 | 0 | 1
  Potassium (mEq/L) >1.1x ULN | 2 | 3 | 0 | 1 | 1
  Chloride (mEq/L) <0.9x LLN | 0 | 1 | 0 | 0 | 0
  Calcium (mg/dL) <0.9x LLN | 0 | 0 | 0 | 0 | 1
  Bicarbonate (mEq/L) <0.9x LLN | 4 | 2 | 0 | 3 | 2
  Creatine Kinase (U/L) >2.0x ULN | 4 | 7 | 1 | 10 | 9
  Troponin I (nanogram per milliliter [ng/mL]) >1.0x ULN | 2 | 3 | 2 | 4 | 4
  Glucose -FASTING (mg/dL) >1.5x ULN | 3 | 5 | 10 | 10 | 2
  Triglycerides -FASTING (mg/dL) >1.3x ULN: number analyzed (Participants) | 94 | 71 | 73 | 100 | 91
  Triglycerides -FASTING (mg/dL) >1.3x ULN | 9 | 7 | 4 | 7 | 5
  Apolipoprotein A1 (mg/dL) >1.5x ULN: number analyzed (Participants) | 93 | 68 | 66 | 93 | 87
  Apolipoprotein A1 (mg/dL) >1.5x ULN | 0 | 1 | 0 | 0 | 0
  Apolipoprotein B (mg/dL) >1.5x ULN: number analyzed (Participants) | 93 | 68 | 66 | 93 | 87
  Apolipoprotein B (mg/dL) >1.5x ULN | 0 | 1 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Change From Baseline in Vital Signs Data Meeting the Pre-defined Categorical Summarization Criteria
Description: Abnormality in change from BL in vital signs included: sitting/semi-supine diastolic blood pressure (BP) increase and decrease from BL of >=20mmHg, systolic BP increase and decrease from BL of >=30mmHg
Time Frame: From BL to Week 28
Population: The safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants with evaluable vital signs data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 11mg MR | PF-06651600 100mg | PF-06650833 400mg MR | PF-06650833 400mg MR + Tofacitinib 11mg MR | PF-06650833 400mg MR + PF-06651600 100mg
Number analyzed (Participants) | 101 | 77 | 77 | 102 | 101
Participants
  Diastolic BP increase >=20mmHg | 1 | 2 | 3 | 6 | 3
  Diastolic BP decrease >=20mmHg | 0 | 0 | 0 | 0 | 0
  Systolic BP increase >=30mmHg | 1 | 3 | 4 | 2 | 3
  Systolic BP decrease >=30mmHg | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Adverse Events of Special Interest
Description: These AEs included severe and opportunistic infection AEs; herpes virus infection AEs; clinically significant categorical increases in hepatic enzymes AST, and ALT and total bilirubin, and potential cases meeting Hy's Law criteria for increased risk of drug induced liver injury (DILI); major adverse cardiovascular events, including pulmonary embolism and deep vein thrombosis, cerebrovascular accident; AEs for decreased renal function, acute kidney injury, clinically significant increases in serum creatinine (Scr) and decreases in estimated glomerular filtration rate (eGFR). Only participants with AEs mentioned above were reported in the table below.
Time Frame: From first dose of study intervention (Day 1) to Week 28
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 11mg MR | PF-06651600 100mg | PF-06650833 400mg MR | PF-06650833 400mg MR + Tofacitinib 11mg MR | PF-06650833 400mg MR + PF-06651600 100mg
Number analyzed (Participants) | 102 | 77 | 77 | 103 | 101
Participants
  Herpes Zoster | 1 | 1 | 0 | 2 | 0
  Oral Herpes | 1 | 0 | 0 | 1 | 2
  ALT Increased | 0 | 0 | 3 | 2 | 0
  AST Increased | 0 | 0 | 2 | 2 | 0
  Hyperbilirubinaemia | 1 | 0 | 0 | 0 | 0
  Transaminases Increased | 0 | 0 | 1 | 0 | 0
  Hepatic Enzyme Increased | 0 | 0 | 1 | 0 | 0
  Liver Injury | 0 | 0 | 1 | 0 | 0

7. Secondary Outcome: Change From Baseline in DAS28-CRP at Week 24
Description: DAS28 is a measure based on assessment of 28 joints for tenderness and swelling (tender and swollen joint counts). DAS28-CRP is derived using differential weighting given to 4 components: tender joint count (range: 0-28), swollen joint count (range: 0-28), patient global assessment (recorded on a visual analog scale [VAS] scale of 0-100 mm), and CRP (milligram per liter). DAS28-CRP score ranges from 0 to 9.4. The lower the DAS28-CRP score is, the better the participant has response (remission = score<2.6, low disease activity = score≤3.2). A negative value in change from BL indicates an improvement.
Time Frame: BL (defined as the last non-missing measurement collected prior to the first administration of study drug on Day 1), Week 24
Population: This endpoint used mITT data set, which included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the randomized intervention. Participants with non-missing data at a given visit were included.
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | PF-06650833 400mg MR + Tofacitinib 11mg MR | PF-06650833 400mg MR + PF-06651600 100mg | Tofacitinib 11mg MR | PF-06651600 100mg | PF-06650833 400mg MR
Number analyzed (Participants) | 84 | 73 | 80 | 54 | 49
Units on a scale | -3.05 [-3.26 to -2.85] | -2.87 [-3.08 to -2.65] | -2.66 [-2.88 to -2.45] | -2.53 [-2.78 to -2.28] | -2.26 [-2.51 to -2.00]

8. Secondary Outcome: American College of Rheumatology (ACR)20, ACR 50, ACR 70, and ACR 90 Responder Rates at Week 12 and Week 24
Description: The American College of Rheumatology's definition for calculating improvement in rheumatoid arthritis (ACR20) is calculated as a >=20% improvement in tender and swollen joint counts and 20% improvement in 3 of the 5 remaining ACR core set measures: patient and physician global assessments, pain, disability, and CRP. Similarly, ACR50, ACR70, and ACR 90 were calculated with the respective percent improvement. Responder rate = number of responders (who had ACR20/50/70/90 response)/(number of responders + non-responders + non-responder assigned by non-responder imputation [NRI] after removal of missingness due to COVID-19 and missing components at a given visit)
Time Frame: BL (defined as the last non-missing measurement collected prior to the first administration of study drug on Day 1), Week 12, Week 24
Population: This endpoint used NRI data set included responders, non-responders, and non-responder assigned by NRI after removal of missingness due to COVID-19 and missing components at a given visit.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Groups:
- PF-06650833 400mg MR: Participants who received PF-06650833 400mg
Arm/Group | PF-06650833 400mg MR + Tofacitinib 11mg MR | PF-06650833 400mg MR + PF-06651600 100mg | Tofacitinib 11mg MR | PF-06651600 100mg | PF-06650833 400mg MR
Number analyzed (Participants) | 103 | 101 | 101 | 77 | 76
Percentage of participants
  ACR20 (Week 12) | 86.41 [79.94 to 91.59] | 79.21 [71.99 to 85.62] | 83.17 [75.94 to 88.98] | 72.73 [63.80 to 80.94] | 75.00 [66.26 to 82.24]
  ACR50 (Week 12): number analyzed (Participants) | 102 | 101 | 101 | 77 | 76
  ACR50 (Week 12) | 62.75 [54.69 to 70.75] | 54.46 [45.79 to 62.57] | 46.53 [38.04 to 55.19] | 44.16 [34.59 to 54.16] | 38.16 [29.16 to 47.81]
  ACR70 (Week 12) | 21.36 [15.35 to 28.95] | 25.74 [19.17 to 33.29] | 23.76 [16.96 to 31.42] | 18.18 [11.34 to 26.08] | 10.53 [5.39 to 18.17]
  ACR90 (Week 12) | 2.91 [1.07 to 6.86] | 3.96 [1.74 to 8.58] | 0.99 [0.10 to 4.12] | 1.30 [0.14 to 5.32] | 1.32 [0.14 to 5.39]
  ACR20 (Week 24): number analyzed (Participants) | 103 | 100 | 101 | 77 | 76
  ACR20 (Week 24) | 75.73 [68.31 to 82.41] | 70.00 [61.87 to 77.31] | 75.25 [67.64 to 82.11] | 67.53 [57.99 to 76.32] | 55.26 [45.20 to 65.01]
  ACR50 (Week 24): number analyzed (Participants) | 103 | 100 | 101 | 77 | 76
  ACR50 (Week 24) | 65.05 [57.08 to 72.34] | 65.00 [56.68 to 72.92] | 65.35 [57.14 to 73.21] | 54.55 [44.56 to 63.80] | 43.42 [33.74 to 53.50]
  ACR70 (Week 24): number analyzed (Participants) | 103 | 100 | 101 | 77 | 76
  ACR70 (Week 24) | 45.63 [37.25 to 54.20] | 44.00 [35.61 to 52.72] | 44.55 [36.60 to 53.22] | 31.17 [22.51 to 40.74] | 27.63 [19.32 to 36.52]
  ACR90 (Week 24): number analyzed (Participants) | 103 | 100 | 101 | 77 | 76
  ACR90 (Week 24) | 12.62 [8.05 to 19.19] | 18.00 [12.27 to 25.23] | 9.90 [5.58 to 16.09] | 5.19 [2.28 to 11.34] | 1.32 [0.14 to 5.39]

9. Secondary Outcome: Change From Baseline in the Tender/Painful and Swollen Joint Count at Week 12 and Week 24
Description: The endpoint included Tender/Painful Joint Count 68 (TJC68) and 28 (TJC28). TJC68 was assessed by a blinded joint assessor to determine the number of joints that were considered tender or painful in upper body and upper/lower extremity. The response to pressure/motion on each joint was assessed using the following scale: Present/Absent/Not Done/Not Applicable (to be used for artificial or missing joints). The 28-joints set is the subset of 68 joints set including the following joints: shoulders, elbows, wrists, metacarpophalangeal joints, proximal interphalangeal joints, and knees. TJC28 was calculated by Pfizer from TJC68. Higher scores indicate higher level of disability.
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Least Squares Mean (90% Confidence Interval); unit: Joints
Arm/Group | PF-06650833 400mg MR + Tofacitinib 11mg MR | PF-06650833 400mg MR + PF-06651600 100mg | Tofacitinib 11mg MR | PF-06651600 100mg | PF-06650833 400mg MR
Number analyzed (Participants) | 100 | 93 | 96 | 69 | 72
Joints
  TJC28 (Week 12) | -9.87 [-10.65 to -9.09] | -9.78 [-10.58 to -8.98] | -9.84 [-10.63 to -9.05] | -9.83 [-10.76 to -8.91] | -8.82 [-9.73 to -7.92]
  TJC68 (Week 12) | -14.96 [-16.09 to -13.83] | -15.66 [-16.81 to -14.50] | -15.32 [-16.47 to -14.18] | -14.80 [-16.13 to -13.46] | -13.76 [-15.07 to -12.46]
  SJC28 (Week 12) | -8.61 [-9.16 to -8.06] | -8.16 [-8.73 to -7.60] | -7.86 [-8.41 to -7.30] | -8.30 [-8.95 to -7.65] | -7.80 [-8.44 to -7.15]
  SJC66 (Week 12) | -11.29 [-11.99 to -10.59] | -10.90 [-11.62 to -10.19] | -10.34 [-11.05 to -9.63] | -10.75 [-11.58 to -9.92] | -10.18 [-11.00 to -9.37]
  TJC28 (Week 24): number analyzed (Participants) | 84 | 74 | 81 | 55 | 49
  TJC28 (Week 24) | -11.33 [-12.06 to -10.61] | -11.44 [-12.20 to -10.68] | -10.60 [-11.34 to -9.86] | -10.47 [-11.34 to -9.59] | -10.31 [-11.20 to -9.42]
  TJC68 (Week 24): number analyzed (Participants) | 84 | 74 | 81 | 55 | 49
  TJC68 (Week 24) | -16.68 [-17.78 to -15.57] | -17.68 [-18.82 to -16.53] | -16.76 [-17.88 to -15.64] | -16.69 [-18.02 to -15.36] | -15.79 [-17.13 to -14.46]
  SJC28 (Week 24): number analyzed (Participants) | 84 | 74 | 81 | 55 | 49
  SJC28 (Week 24) | -8.83 [-9.34 to -8.31] | -9.44 [-9.98 to -8.90] | -8.76 [-9.29 to -8.24] | -8.71 [-9.33 to -8.08] | -8.28 [-8.92 to -7.65]
  SJC66 (Week 24): number analyzed (Participants) | 84 | 74 | 81 | 55 | 49
  SJC66 (Week 24) | -11.41 [-12.02 to -10.80] | -12.38 [-13.03 to -11.74] | -11.59 [-12.21 to -10.97] | -11.45 [-12.19 to -10.71] | -11.10 [-11.86 to -10.34]

10. Secondary Outcome: Change From Baseline in the Physician's Global Assessment (PhGA) of Arthritis at Week 12 and Week 24
Description: PhGA of Arthritis is an evaluation done by investigator based on the participant's disease signs, functional capacity and physical examination, and should be independent of the Patient's Global Assessment of Arthritis. The investigator's response was recorded using a 100 mm VAS. Physician's Global Assessment score ranges from 0 to 100. Higher scores indicate higher level of disability. A negative value in change from BL indicates an improvement.
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | PF-06650833 400mg MR + Tofacitinib 11mg MR | PF-06650833 400mg MR + PF-06651600 100mg | Tofacitinib 11mg MR | PF-06651600 100mg | PF-06650833 400mg MR
Number analyzed (Participants) | 100 | 93 | 96 | 69 | 72
Units on a scale
  PhGA of Arthritis (Week 12) | -43.50 [-46.32 to -40.69] | -41.20 [-44.06 to -38.34] | -40.86 [-43.72 to -38.00] | -38.62 [-41.95 to -35.28] | -31.56 [-34.82 to -28.30]
  PhGA of Arthritis (Week 24): number analyzed (Participants) | 84 | 74 | 81 | 55 | 49
  PhGA of Arthritis (Week 24) | -47.50 [-50.13 to -44.87] | -48.21 [-50.95 to -45.47] | -47.31 [-49.98 to -44.63] | -43.42 [-46.60 to -40.25] | -39.27 [-42.49 to -36.05]

ADVERSE EVENTS:
Time Frame: From first dose of study intervention (Day 1) to Week 28
Description: SAEs and non-serious AEs were recorded on the case report form. SAEs were also reported on the Clinical Trial SAE report form to Pfizer Safety within 24 hours of awareness. The same event may appear as both an AE and SAE. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs/AEs.
Groups:
- PF-06650833 400mg MR: Participants received PF-06650833 400mg MR tablets QD.
Arm/Group | Tofacitinib 11mg MR | PF-06651600 100mg | PF-06650833 400mg MR | PF-06650833 400mg MR + Tofacitinib 11mg MR | PF-06650833 400mg MR + PF-06651600 100mg
All-Cause Mortality (participants affected / at risk) | 1/102 | 0/77 | 0/77 | 0/103 | 0/101
Serious Adverse Events (participants affected / at risk) | 3/102 | 3/77 | 3/77 | 0/103 | 1/101
Other Adverse Events (participants affected / at risk) | 24/102 | 18/77 | 11/77 | 19/103 | 26/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib 11mg MR (N=102) | PF-06651600 100mg (N=77) | PF-06650833 400mg MR (N=77) | PF-06650833 400mg MR + Tofacitinib 11mg MR (N=103) | PF-06650833 400mg MR + PF-06651600 100mg (N=101)
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Coronavirus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin squamous cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib 11mg MR (N=102) | PF-06651600 100mg (N=77) | PF-06650833 400mg MR (N=77) | PF-06650833 400mg MR + Tofacitinib 11mg MR (N=103) | PF-06650833 400mg MR + PF-06651600 100mg (N=101)
Nausea (Gastrointestinal disorders) | 4 | 5 | 2 | 1 | 3
Nasopharyngitis (Infections and infestations) | 3 | 2 | 1 | 3 | 6
Urinary tract infection (Infections and infestations) | 5 | 1 | 1 | 7 | 3
SARS-CoV-2 test positive (Investigations) | 7 | 1 | 2 | 4 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 5 | 1 | 2 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 | 4 | 4 | 1 | 1
Headache (Nervous system disorders) | 4 | 4 | 2 | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-02-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT04413617/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT04413617/SAP_001.pdf